CLINICAL TRIAL: NCT06072027
Title: Evaluation of the Real-life Contribution of VISIOCYT Bladder Cytology in Patients With Suspected Bladder Tumor or in the Follow-up of a Bladder Tumor
Brief Title: Evaluation of VISIOCYT Bladder Cytology in Real Life
Acronym: VISIOCYT2
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: VISIOCYT2-IPC 2020-072
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will be offered to all consecutive patients undergoing scheduled cystoscopy at the Hospitalisation De Jour (HDJ) Chirurgicale, either as part of a diagnostic approach in the event of suspected bladder tumor (exploration of macroscopic hematuria in particular), or as part of the follow-up of a bladder tumor, according to current recommendations (French ccAFU guidelines - update 2020-2022: bladder cancer).

Once non-opposition has been obtained, clinical data at the time of inclusion will be collected and pseudonymized. Urine is collected prior to cystoscopy, on voided urine, for a minimum sufficient quantity of 50 ml. The urine sample is then separated into transport jars, one of which is used for standard cytological analysis, the other for VISIOCYT cytology (sent to a laboratory platform).

In the event of a tumor or suspicious lesion detected at the cystoscopy, a trans-urethral bladder resection (TURB) will be scheduled. Anatomopathological data from this RTUV will also be collected for comparative analysis to establish the diagnostic performance of the test.

The tests performed (apart from the urine sample) are part of the usual care pathway. No additional visits will be specifically requested by the protocol. Data from examinations carried out as part of standard pathology management, or suspected pathology, will be used for this research.

At the same time, prospective questionnaires on patients' preferences with regard to the various diagnostic examinations for bladder tumours (discrete choice analysis) will be given to patients and completed at the time of cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age,
* Signed consent to participate,
* Affiliation with a social security scheme, or beneficiary of such a scheme,
* Patient to undergo cystoscopy for diagnosis (suspected bladder tumor) or follow-up of bladder tumor

Exclusion Criteria:

* Patients managed or followed up for a bladder tumor of non-urothelial histology,
* Renal transplant patients,
* Patient having received pelvic radiotherapy,
* Pregnant or potentially pregnant women (of childbearing age, without effective contraception) or nursing mothers,
* Person in an emergency situation, adult under legal protection (guardianship, curatorship or safeguard of justice), or unable to express consent,
* Inability to undergo medical follow-up for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient to undergo cystoscopy for diagnosis (suspected bladder tumor) or follow-up of bladder tumor
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-06-09 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
negative predictive value | 1 day
  negative predictive value of the VisioCyt® Bladder test. The second primary endpoint was the sensitivity of the VisioCyt® Bladder test.

SECONDARY OUTCOMES:
Diagnostic performance - VisioCyt® Bladder test | 1 day
  Diagnostic performance of different algorithmic versions (V1 Versus V2) of the VisioCyt® Bladder ® test (sensitivity, specificity, positive predictive value, negative predictive value)
Diagnostic performance - standard cytology | 1 day
  Diagnostic performance of standard cytology (sensitivity, specificity, positive predictive value, negative predictive value)
Diagnostic performance of cystoscopy | 1 day
  Diagnostic performance of cystoscopy (sensitivity, specificity, positive predictive value, negative predictive value)
Patient preference | 1 day
  Patient preference for different diagnostic tests (discrete choices)

CONTACTS AND LOCATIONS:
Overall Officials: Jihane PAKRADOUNI, PharmD, Study Director — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France